CLINICAL TRIAL: NCT04157829
Title: Evaluation of the Performance and Safety of a Scintillating Lamp Developed to Improve the Reading of Dyslexic Patients
Brief Title: Evaluation of the Performance and Safety of a Medical Device Developed to Improve the Reading of Dyslexic Patients
Acronym: DysLight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SATT Ouest Valorisation (Other)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DysLight
Record Dates: First submitted 2019-11-04; First posted 2019-11-08 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Dyslexia
Keywords: Dyslexia; Reading disorder
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scintilling lamp- Classic lamp (Experimental)
  Interventions: Device: Scintilling lamp; Device: Classic lamp
- Classic lamp- Scintilling lamp (Experimental)
  Interventions: Device: Scintilling lamp; Device: Classic lamp

INTERVENTIONS:
Device: Scintilling lamp — Lamp with a standardized scintilling
Device: Classic lamp — Lamp without a scintilling

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of a new medical device on the improvement of reading skills of dyslexic patients.

DETAILED DESCRIPTION:
Dyslexia is defined as a specific learning disability that is characterized by reading difficulties, in the absence of intellectual disability, neurological or psychiatric disorder, uncorrected sensory disturbance (sight, hearing) or an educational deficiency.

Dyslexia appears in the child from the earliest stages of learning in the form of a difficulty in mastering the learning of reading. This disorder is manifested by a generally hesitant reading, slowed down, full of errors, requiring a lot of effort for the child and may impact his reading comprehension. The dyslexia-related deficiency is of variable intensity depending on the individual; it may be accompanied by calculus disorders (dyscalculia), oral language (dysphasia), motor coordination (dyspraxia) or attention disorders with or without hyperactivity. In nearly 40% of cases, a child affected by Dys disorders presents several learning disorders.

To date, the causes of dyslexia are not yet clearly established. The wide variety of symptoms and disorders associated with dyslexia does not facilitate the identification of precise neurobiological / psycho cognitive mechanisms. There are therefore several theories: phonological, visual, temporal, cerebellar or proprioceptive auditory processing.

Recently, following work published in 2017, an anatomical cause based on Maxwell's spots could also be a cause of dyslexia.

The aim of this study is to evaluate a new medical device to compensate this probable anatomical cause.

ELIGIBILITY:
Inclusion Criteria:

* Schooled in CE2, CM1 or CM2,
* French mother tongue,
* For whom developmental dyslexia has been diagnosed by a health professional who specializes in this learning disorder,
* Presenting an IQ ≥ 80 and ≤130 according to the WISC-V test performed by a psychologist,
* For which a written consent was obtained regarding his study participation.

Exclusion Criteria:

* With medical history or presenting a neurological pathology,
* Presenting a developmental disorder (autism, ADHD, ...),
* Presenting hearing disorders,
* Presenting visual disorders,
* Any other condition that, in the opinion of health professionals, could impair its ability to complete the study or could pose a significant risk.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Reading performance aloud of a text with french E.L.FE Test | 1 day
  E.L.FE Test (=Evaluation de la Lecture en FluencE) - "Monsieur Petit" and "Le Géant égoïste" texts : percentile

SECONDARY OUTCOMES:
Reading performance aloud of isolated words with french BALE Test | 1 day
  BALE test (=Batterie Analytique de Langage Ecrit): percentile
Security: incidence of Adverse Events | 1 day
  By questioning the patient & the speech therapist - evaluation of adverse effects due to scintilling lamp (Yes/ No): headache, nausea, dizziness, fatigue and eye fatigue. Accotding to patient questioning and clinical exam, the Adverse Event Table will be completed (description, dates, severity, imputability, action,...).
Patient's satisfaction regarding reading fluency | 1 day
  patient interview with VAS (Visual Analogue Scale): 0 - 100 mm
Speech therapist's satisfaction regarding Securirty, Performance and usability of scintilling lamp | 1 day
  speech therapist interview with 4 points - Likert scale (Very good, Good, Moderate, Bad)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Allaire, Dr, Principal Investigator — CHU Rennes
Locations (4):
- France (4):
  - Dr Laurence Derieux, Caen
  - Dr Luc-Marie Virlet, Faumont
  - Dr Hugo Peyre, Paris
  - Dr Catherine ALLAIRE, Rennes